CLINICAL TRIAL: NCT01705678
Title: An Investigation Into the Effects of Krill Oil vs. Fish Oil on Markers of Cardiovascular Disease in Males With Metabolic Syndrome
Brief Title: Investigation Into the Effects of Krill Oil vs. Fish Oil on Markers of Cardiovascular Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Responsible Party: Principal Investigator, Ian G. Davies, Dr Ian G. Davies, Liverpool John Moores University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: KO-001
Record Dates: First submitted 2012-04-12; First posted 2012-10-12 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Metabolic Syndrome
Keywords: Males; Metabolic syndrome; Otherwise healthy
MeSH Terms: conditions — Metabolic Syndrome | interventions — Fish Oils

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Krill oil (Active Comparator): Krill oil will be compared to fish oil as an active comparator
  Interventions: Dietary Supplement: Fish oil
- Fish oil (Active Comparator): Fish oil 500 mg of DHA/EPA
  Interventions: Dietary Supplement: Krill oil

INTERVENTIONS:
Dietary Supplement: Krill oil — Krill oil 300 mg DHA/EPA daily for 6 weeks
  Arms: Fish oil
Dietary Supplement: Fish oil — Fish oil 500 mg DHA/EPA daily for 6 weeks
  Arms: Krill oil

SUMMARY:
There is some evidence that dietary supplementation with fish oil has health benefits, especially in respect of some of the known risk factors for cardiovascular (heart) disease such as cardiac arrhythmia. However, supplies of fish oil are limited, and it is desirable to validate alternative sustainable sources of the important omega-3 fatty acid components. It has been suggested that oil from krill, which are small marine crustaceans, may be as effective or possibly more beneficial than fish oil, and may provide a more effective and beneficial supplement. Dietary management of cardiovascular health parameters (such as blood lipids)is becoming more and more important as the rising trends in obesity nationally and worldwide are leading to escalating incidence of diabetes and heart disease. The investigators propose to use some specific novel lipid measurements of cardiovascular risk to test this possibility in a group of men who, although generally healthy, show some risk factors in terms of their weight and metabolic profile.This pilot study will provide preliminary data to show whether krill oil has similar or different effects from fish oil on the cardiovascular health of overweight but otherwise healthy men, and in particular will provide detailed information on alterations in novel lipid markers of cardiovascular disease, which may be a better diagnostic tool than classical lipid measurements (e.g. serum cholesterol). The investigators have been developing and validating new techniques to measure emerging lipid markers of cardiovascular risk accurately and will continue to develop and investigate these techniques during the course of this project. The investigators hypothesise that krill oil will be more efficacious in reducing markers of risk relating to cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* waist circumference ≥ 94cm

Plus any two of the below:

* Raised triglycerides : ≥ 150 mg/dL (1.7 mmol/L)
* Reduced HDL cholesterol: < 40 mg/dL (1.03 mmol/L)
* Raised blood pressure: ≥ 130/85 mm Hg
* Raised fasting plasma glucose: ≥ 100 mg/dL (5.6 mmol/L)

Exclusion Criteria:

* Drug treatment for cardiovascular disease or diabetes,
* currently taking fish oil supplements
* Individuals who would require carers or guardians to make decisions
* Known history of liver disease

Ages: 35 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-05; Primary Completion 2010-09 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Change in Plasma Triglycerides at 3 weeks | Change from baseline at 3 weeks
  Change in plasma triglycerides from baseline to midpoint
Change in plasma high density lipoprotein cholesterol at 3 weeks | Change from baseline at 3 weeks
  Change in plasma High density lipoprotein cholesterol from baseline to midpoint
Change in plasma glucose at 3 weeks | Change from baseline at 3 weeks
  Change in plasma glucose from baseline to midpoint
Change in waist circumference | Change from baseline at 6 weeks
  Change in waist circumference from baseline to endpoint
Change in systolic blood pressure | Change from baseline at 6 weeks
  Change in systolic blood pressure from baseline to endpoint
Change in Diastolic blood pressure | Change from baseline at 6 weeks
  Change in diastolic blood pressure from baseline to endpoint
Change in plasma triglycerides at 6 weeks | Change from baseline at 6 weeks
  Change in plasma triglycerides at baseline to endpoint
Change in plasma glucose at 6 weeks | Change from baseline at 6 weeks
  Change in plasma glucose from baseline to endpoint
Change from baseline high density lipoprotein cholesterol at 6 weeks | Change from baseline at 6 weeks
  Change in high density lipoprotein cholesterol from baseline to endpoint

SECONDARY OUTCOMES:
Change in Body mass | Change from baseline at 6 weeks
  Change in body mass measured at baseline to endpoint
Change in plasma total cholesterol | Change from baseline at 3 weeks
  Change in plasma cholesterol from baseline to midpoint
Change in body mass index | Change from baseline at 6 weeks
  Change in body mass index at baseline to endpoint
Change in plasma cholesterol at 6 weeks | Change from baseline at 6 weeks
  Change in plasma cholesterol from baseline to endpoint
Change in plasma insulin at 3 weeks | Change from baseline at 3 weeks
  Change in plasma insulin from baseline to midpoint
Change in plasma insulin at 6 weeks | Change from baseline at 6 weeks
  Change in plasma insulin from baseline to endpoint
Change in small, dense low density lipoprotein cholesterol at 6 weeks | Change from baseline at 6 weeks
  Change in small, dense low density lipoprotein cholesterol from baseline to endpoint
Change in plasma low density lipoprotein cholesterol at 3 weeks | Change from baseline at 3 weeks
  Change in plasma low density lipoprotein cholesterol from baseline to midpoint
Change in plasma low density lipoprotein cholesterol at 6 weeks | Change from baseline at 6 weeks
  Change in plasma low density lipoprotein cholesterol from baseline to endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Ian G Davies, PhD, Principal Investigator — Liverpool John Moores University